CLINICAL TRIAL: NCT03940287
Title: Efficacy of Muscle Energy Technique and Kinesiotape Application in Addition to Other Physiotherapeutic Intervention in Patients With Mechanical Sacroiliac Joint Dysfunction
Brief Title: Muscle Energy Technique and Kinesiotaping in Mechanical Sacroiliac Joint Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 lockdown
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Supervisor and Associate Professor, Department of Pediatric and Neonatal Physiotherapy, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMDU/IEC/1370; U1111-1232-1305 (Other: UTN by WHO International Clinical Trial Registry Platform)
Record Dates: First submitted 2019-05-01; First posted 2019-05-07 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: Sacroiliac Joint pain; Low back pain; Pelvic girdle pain
MeSH Terms: conditions — Low Back Pain; Pelvic Girdle Pain

STUDY DESIGN:
Intervention Model Description: Two group pre test post test Randomized Clinical Design
Who Masked: Participant
Masking Description: Participant blinded (Single blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique and Conventional Physiotherapy (Experimental): Muscle Energy Technique will be given with conventional physiotherapy for 3 days per week and will be continue for 4 weeks, where each session of Muscle Energy Technique will be repeated for 3-5 repetitions.
  Interventions: Other: Muscle Energy Technique; Other: Conventional physiotherapy
- Kinesiotaping and Conventional Physiotherapy (Experimental): Kinesiotape application will be given with conventional physiotherapy for 3 days per week and will be continue for 4 weeks
  Interventions: Other: Kinesiotape application; Other: Conventional physiotherapy

INTERVENTIONS:
Other: Muscle Energy Technique — Muscle energy technique will be given in two different position. For anterior in- nominate rotation and posterior in- nominate rotation patient position will be in supine lying position.
  For weakened muscle,piriformis application the patient should be side-lying position, close to the edge of the table, affected side uppermost, both legs flexed at hip and knee.
  The therapists stand facing the patient at hip level,then patient should be close enough to the edge of the table for the therapist to stabilize the pelvis against his trunk. The angle of hip flexion should not exceed 60°, and then places one hand on the contralateral ASIS to prevent pelvic motion, while the other hand is placed against the lateral flexed knee as this is pushed into resisted abduction to contract piriformis.
  Isometric contraction should be hold for 3-5 second and that particular method will be repeated for 7-10 times.
  Arms: Muscle Energy Technique and Conventional Physiotherapy
Other: Kinesiotape application — Kinesiotaping will be applied to piriformis muscle and Sacroiliac joint (SIJ). This tape will be applied in I shape to both sides of the spine from sacrum to Anterior Superior Iliac Spine. For SIJ taping same 5 cm KT tape will be used, it will be applied from below posterior sacroiliac spine to opposite side. Here patient should be in standing position.
  For Piriformis application patient will be in side lying position where the affected leg will be placed uppermost with hip in flexion, adduction, and internal rotation , then the application will be performed. The base of the tape will be placed over contralateral part of sacrum and then make a Y strip with no tension will be attached over the greater trochanter of femur.
  Arms: Kinesiotaping and Conventional Physiotherapy
Other: Conventional physiotherapy — Hydro-collator pack will be used superior to the affected area for at-least 15 minute to reduce the stiffness. Hydocollator pack will be wrap twice with a thick towel and then it will be placed to the affected part.

SUMMARY:
Background:

Mechanical sacroiliac joint dysfunction is associated with pain and stiffness which can later on gives restriction of overall motion. Total 60% of the body weight is mainly received by the sacroiliac joint and it is related with pelvis and lower extremity. Due to Bio- mechanical alteration muscles around the joint area get weakened.Muscle energy technique helps to improve body's normal function by giving strength as well as decrease pain and stiffness and Kinesiotaping also helps to stabilize the joint structure by giving more functional benefit.

Aim:

The Aim of the study is to evaluate the efficacy of Muscle energy technique & Kinesiotaping in addition to other physio-therapeutic intervention in patients with Mechanical Sacroiliac joint Dysfunction.

Methods:

This study is a randomized clinical trial and subjects will recruit on the basis of inclusion criteria. Age group between 30 to 50 years of mechanical sacroiliac joint dysfunction patients will be taken. Any pathological condition like inflammation of sacroiliac joint and fracture of pelvic bone will be excluded. Patient will be randomized on the basis of SNOSE method. After randomization in two equal group treatment will be given and data will be analyzed separately. One Experimental group will receive Muscle energy technique and conventional physiotherapy and another experimental group will receive Kinesiotaping and conventional physiotherapy. Modified Oswestry Disability Index helps to evaluate functional limitation associated with Mechanical Sacroiliac joint Dysfunction.

Data Analysis:

Normality of the collected data will be established by Shapiro wilk test. Based on the normality, descriptive statistics data will be expressed as mean± standard deviation or median and intra-quartile range. Within group comparison will be calculated by paired-t test or Wilcoxon Signed Rank test and between group comparison will be done through Independent-t test or Mann-Why U test. P value will be set at significance level(0.05).

DETAILED DESCRIPTION:
1. Introduction:

   Mechanical Sacroiliac joint dysfunction (SIJD) is the most common source of low back pain and affects 70-85% adults. It is also associated with groin & buttock pain and sometime also leg pain. Non discogenic pain can also be occur due to dysfunction around Sacroiliac Joint. Sacroiliac joint dysfunction also called as pelvic girdle pain (PGP), which arises from several intra-articular structures, anterior sacroiliac ligament, posterior sacroiliac ligament, articular cartilages. Sacroiliac joint pain is one of the common sources of mechanical low back pain. This may lead to bio-mechanical alteration in structure around pelvis.Where as Muscle Energy Technique(MET) involves physiological response of the antagonists of a muscle which has been isometrically contracted. Mainly MET is a soft tissue manipulation which include force generated by the patient may be maximum muscle contraction are twitch of the muscle. Where as functional stability as well as mobility can be achieved by Kinesiotape application.

   1.1: Problem statement:

   Mainly sacroiliac joint dysfunction associated with altered arthokinematics due to muscle weakness. Kinesiotaping and MET will be helpful if they are used with conventional physiotherapy. Thus there is need to find out the efficacy of MET and Kinesiotaping in addition to conventional physiotherapy in patients with mechanical SIJD.

   1.2:Purpose of the study:

   The purpose of the study is to find out the efficacy of MET and Kinesiotaping in addition to conventional physiotherapy in patients with mechanical sacroiliac joint dysfunction.

   1.3: Objectives of the study:

   1.3.1:To determine the effect of MET and Kinesiotaping in addition to conventional physiotherapy in patients with Mechanical Sacroiliac joint Dysfunction. 1.3.2:To compare the effect of MET &Kinesiotaping in patients with Mechanical Sacroiliac joint dysfunction.
2. Procedure:

The study will be a Two group pre test post test Randomized clinical trial. The study protocol has been approved from the Institutional Ethics Committee of Maharishi Markandeshwar Deemed to be University.

MET Application: MET will be used with conventional treatment in Experimental Group 1. MET will be applied for posterior and anterior in-nominate and for weakened muscles like piriformis.

Here patient will be asked to apply 20% force against therapist force and hold that contraction for 10 seconds with 3-5 repetitions.The treatment will be given for 3 times a week and continued for 4 weeks.

Kinesiotaping will be given with conventional physiotherapy in Experimental Group 2. In this group KT will be applied to piriformis muscle and Sacroiliac joint (SIJ).

For piriformis application patient will be in side lying position where the effected leg will be placed uppermost with hip in flexion, adduction, and internal rotation and Y strips will be used & treatment will be given for 4 weeks with 3 alternative days in a week.

Conventional Physiotherapy will be given in both the groups. Before going for intervention Hydrocollator pack will be given in both the groups for at least 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the low back, buttock and groin area
* Restricted Sacroiliac joint motion as tested by clinical tests (Standing Flexion & Sitting Flexion test)
* Leg pain more than 4 weeks but less than 1 year

Exclusion Criteria:

* Inflammation in sacroiliac joint like sacroilitis
* Pregnancy
* Pelvic bone Fractures
* Metallic implants (endoprostheses) in pelvis
* Malignancy
* Inflammatory bowel disease

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Digitalized Pain Pressure Algometer | 2 weeks
  It is an important tool for measuring pain pressure threshold level
Hand Held Dynamometer | 2 weeks
  It is useful tool for calculating muscle strength of lower extremity

SECONDARY OUTCOMES:
Modified Oswestry Disability Index | 2 weeks
  It is an extremely important tool used to measure a patients permanent functional disability. The total score ranges from 0-50. For each section total possible score is 5.
  0-20%- Minimal disability 20-41%-Moderate disability 41-60%-Severe disability 61-80%-Crippled 81-100%-Bed bound

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Sarkar, BPT, (MPT), Principal Investigator — Department of Musculoskeletal Physiotherapy, MMIPR
Locations (1):
- Maharishi Markandeshwar Hospital, Mullana, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No
It is not yet decided

REFERENCES:
- [Result] Shinde M, Jagtap V. Effect of Muscle Energy Technique and Mulligan Mobilization in Sacroiliac Joint Dysfunction. Glob J Res Anal. 2018;(3):79-81.
- [Result] Society TK, Therapy P, Journal T, Therapy KP, Ther KP, Scholar G, et al. The effects of spinal decompression therapy on pain and disability in patients with chronic low back pain. J Korean Phys Ther. 2017;29(6).